CLINICAL TRIAL: NCT01397500
Title: Growth Hormone and Gonadotropin Deficiency After Brain Injury (Traumatic Brain Injury, Subarachnoidal Hemorrhage, Ischemic Stroke): the Effects of Hormone Replacement on Cognition, Quality of Life and Body Composition
Brief Title: Hormone Treatment in Growth Hormone and Testosterone Deficient Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment problems due to change of patient population at site.
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Collaborators: Schoen Clinic Bad Aibling (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS/Muenchen 02
Record Dates: First submitted 2011-05-17; First posted 2011-07-19 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Hormone Deficiency
MeSH Terms: interventions — Human Growth Hormone; testo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Genotropin (Active Comparator): 6 months Genotropin (open treatment)
  Daily dose:
  Male < 45 years: 0,4 mg; ≥ 45 years: 0,2 mg Female < 45 years: 0,5 mg; ≥ 45 years: 0,3 mg Starting with half of the dose for the first 4 weeks.
  Interventions: Drug: Genotropin
- Testosterone undecannoate (Active Comparator): 18 weeks testosterone undecanoate/placebo (double-blind treatment) 1000 mg/4 ml at baseline and after 6 weeks
  Interventions: Drug: Testosterone undecannoate
- control group (No Intervention): No Intervention.

INTERVENTIONS:
Drug: Genotropin — Genotropin administered sc once a day by patient or caregiver.
  Other Names: GH
  Arms: Genotropin
Drug: Testosterone undecannoate — Testosterone undecannoate administered twice (6 week Interval) im by investigator.
  Other Names: Testo
  Arms: Testosterone undecannoate

SUMMARY:
Growth hormone and gonadotropin deficiency after brain injury (traumatic brain injury, ischemic stroke, subarachnoidal hemorrhage): the effects of hormone replacement on cognition, quality of life and body composition Randomized, controlled, 3 arm (group 2: double-blind; groups 1 and 3: open), multi-center, pilot study (Phase II)

DETAILED DESCRIPTION:
The aim of the study is to investigate the influence of growth-hormone replacement on cognition, quality of life, body mass index, body composition and reorganization of brain activity of hypopituitary patients in a stable, chronic phase after brain injury compared to control patients and the influence of testosterone replacement in gonadotropin deficient patients compared to placebo treated control patients.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

1. Age
2. F/M
3. Stable phase after TBI, SAH or IS
4. Stable substitution of other hormonal axes
5. GH below 6 ng/ml after stimulation with ITT or GH below cut-off in GHRH/arginine test using BMI-adjusted cut-off limits, GHRH/arginine test should be done only in patients denying or with a contraindication for ITT
6. Written informed consent

Group 2:

1. Age
2. M
3. PSA in normal range
4. Stable phase after TBI, SAH or IS
5. Stable substitution of other hormonal axes
6. Below 3.5 ng/ml testosterone
7. Written informed consent

Group 3:

1. Age
2. F/M
3. Stable phase after TBI, SAH or IS
4. GH higher 6 ng/ml after stimulation with ITT or GH below cut-off in GHRH/arginine test using BMI-adjusted cut-off limits, GHRH/arginine test should be done only in patients denying or with a contraindication for ITT
5. Written informed consent

Exclusion Criteria:

Group 1:

1. Pregnancy/lactation period
2. Women of childbearing potential not using an adequate method of birth control
3. Men not willing to use an adequate method of birth control
4. Previous or concomitant medication with GH
5. Hypersensitivity to GH
6. Drug or alcohol abuse
7. Condition which in opinion of investigator makes patient unsuitable for inclusion
8. Participation in another clinical trial with investigational new drug
9. Planned treatment or changes in established treatment with other drug which might significantly influence GH axis or cognitive function
10. Non-ability to perform testing
11. Presence of other conditions listed in contraindications or warnings in local SPC of GH
12. Onset of GH-deficiency before BI

Group 2:

1. Men not willing to use an adequate method of birth control
2. Previous or concomitant medication with androgens or anabolic steroids within 12 months
3. Hypersensitivity to active substances or excipients of Nebido®
4. Drug or alcohol abuse
5. Condition which in opinion of investigator makes patient unsuitable for inclusion
6. Participation in another clinical trial with investigational new drug
7. Planned treatment or changes in established treatment with other drug which might influence gonadotrophic axis or cognitive function
8. Severe disturbances in articulation, visual faculty, hearing
9. Presence of other conditions listed in contraindications or warnings in local SPC of Nebido®
10. Onset of hormonal deficiency before BI
11. Suspicion or known history of prostate or breast cancer or other hormone dependent neo plasia as well as history of malignancy within last 5 years
12. Abnormal finding on DRE
13. PSA higher 4 ng/ml
14. History of clinically significant post void residual urine before BI
15. Suspicion or known history of liver tumor
16. Blood coagulation irregularities presenting an increased risk of bleeding after i.m injections
17. Hypercalcemia accompanying malignant tumors
18. Sleep apnea
19. Polycythemia
20. Haematocrit higher than 50 %
21. Concurrent use of DHEA, anabolic steroids, clomipramine, antiandrogens, estrogen, ACTH, corticosteroids, oxyphenbutazone
22. Uncontrolled thyroid disorders like diabetes mellitus, epilepsia, migraine, hypertension, coronary heart disease as well as hepatic, renal or cardiac insufficiency
23. Patients requiring or undergoing fertility treatment
24. Condition which in opinion of investigator makes patient unsuitable for inclusion
25. Non-ability to perform cognitive testing
26. Onset of androgen deficiency before BI.

Group 3:

1. Previous or concomitant medication with androgens, GH or anabolic steroids within 12 months
2. Drug or alcohol abuse
3. Condition which in opinion of investigator makes patient unsuitable for inclusion
4. Participation in another clinical trial with investigational new drug
5. Planned treatment or changes in established treatment with other drug which might influence gonadotrophic axis or cognitive function
6. Severe disturbances in articulation, visual faculty, hearing
7. Non-ability to perform cognitive testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months
  Quality of Life (QoL) was measured with the following questionnaires prior to treatment and after treatment:
  * SF-12 short-form health questionnaire (12 items, score: min. 12/max. 47)
  * QoL-AGHDA Assessment of GHD in Adults (25 items: yes/no answers)
  * EQ-5 D Euroquol (5 items, scale per items from 1 (no problems) to 3 (severe problems); 1 Likert scale (0 worst-100 best) to measure health status)
  * BDI Beck Depression Inventory (21 items, score: min. 0/max. 63)
  * PSQI Pittsburgh Sleep Quality Index: (4 items regarding sleep duration, 11 items regarding sleep quality, 1 item regarding sleeping medication, 2 item regarding daytime dysfunction, 1 item regarding sleeping habit; 5 items for third-party assessment)
  * QOLIBRI Quality of Life after Brain Injury (37 items, scale per item from 1 (not at all) to 5 (very much) QoL was measured with difference between mean scores of the respective questionnaires, determined before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Sievers, MD, Principal Investigator — Max Planck Institute
Locations (1):
- Max Planck Institute, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Leonhardt M, Kopczak A, Schapers B, Limbrock J, Samann PG, Czisch M, von Steinbuechel N, Jordan M, Schneider HJ, Schneider M, Sievers C, Stalla GK. Low Prevalence of Isolated Growth Hormone Deficiency in Patients After Brain Injury: Results From a Phase II Pilot Study. Front Endocrinol (Lausanne). 2018 Dec 17;9:723. doi: 10.3389/fendo.2018.00723. eCollection 2018. PMID 30619080